CLINICAL TRIAL: NCT03951597
Title: a Single-arm Study of Combined Therapy Using Oxaliplatin and Gemcitabine Chemotherapy, Lenvatinib and Programmed Cell Death Protein 1 Antibody (JS001) for Patients With Advanced and Unresectable Intrahepatic Cholangiocarcinoma
Brief Title: Combined Therapy Using Oxaliplatin and Gemcitabine Chemotherapy, Lenvatinib and PD1 Antibody (JS001) for Patients With Advanced and Unresectable Intrahepatic Cholangiocarcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: zs-ICC-2019
Record Dates: First submitted 2019-05-14; First posted 2019-05-15 (Actual); Last update posted 2021-07-07 (Actual); Status verified 2021-07

CONDITIONS: Cholangiocarcinoma, Intrahepatic
Keywords: intrahepatic cholangiocarcinoma; oxaliplatin and gemcitabine chemotherapy; Lenvatinib; programmed cell death protein 1 antibody
MeSH Terms: conditions — Cholangiocarcinoma | interventions — lenvatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Combined therapy using Gemox, Lenvatinib and PD1 (Experimental): 1. Gemox chemotherapy Day1 oxaliplatin 85mg/m2+ gemcitabine 1g/m2, Day8 gemcitabine 1g/m2 Three weeks is a course of treatment with a total of 6 courses.
  2. Lenvatinib (8mg/d), continuous use for 1 year.
  3. PD-1 antibody (JS001) (240mg every 3 weeks), continuous use for 1 year.
  Interventions: Drug: combined therapy using oxaliplatin and gemcitabine chemotherapy, Lenvatinib and PD1 antibody (JS001)

INTERVENTIONS:
Drug: combined therapy using oxaliplatin and gemcitabine chemotherapy, Lenvatinib and PD1 antibody (JS001) — 1. Gemox chemotherapy Day1 oxaliplatin 85mg/m2+ gemcitabine 1g/m2, Day8 gemcitabine 1g/m2 Three weeks is a course of treatment with a total of 6 courses.
  2. Lenvatinib (8mg/d), continuous use for 1 year.
  3. PD-1 antibody (JS001) (240mg every 3 weeks), continuous use for 1 year.

SUMMARY:
In this phase 2 study, the investigators aim to evaluate the effects and safety of combined therapy using oxaliplatin and gemcitabine chemotherapy, Lenvatinib and immune checkpoint inhibitor PD-1 antibody (JS001) for patients with advanced and unresectable intrahepatic cholangiocarcinoma

DETAILED DESCRIPTION:
Most intrahepatic cholangiocarcinoma (ICC) patients are often accompanied by local or distant metastases and lose the opportunity for surgical resection. For patients with unresectable ICC who have been in stages IIIb and IV (AJCC/UICC, V2, 2018), the survival time is less than 4 months, and there is currently no standard treatment. The Gemox chemotherapy (oxaliplatin + gemcitabine) has been used in the treatment of advanced intrahepatic cholangiocarcinoma, but the efficacy is still unsatisfactory. Lenvatinib is a small molecule multi-kinase inhibitor, the main targets including VEGFR1-3, fibroblast growth factor receptor 1-4, PDGFRα, RET(ret proto-oncogene ), KIT(KIT proto-oncogene, receptor tyrosine kinase), have anti-angiogenic effects, have been proven effective in hepatocellular carcinoma. In recent years, monoclonal antibodies against programmed cell death protein 1 (PD1) have shown remarkable therapeutic effects in the treatment of various solid tumors. Combined with other means such as chemotherapy and targeted drugs is an important direction to improve the therapeutic effect of immunological checkpoint inhibitors. In this study, the investigators aim to evaluate the effects and safety of Gemox chemotherapy combined with Lenvatinib and immune checkpoint inhibitor PD-1 antibody (JS001) for patients with advanced and unresectable intrahepatic cholangiocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. The patient must be required to sign an informed consent form;
2. age 18-75 years old, male or female;
3. Eastern Cooperative Oncology Group (ECOG) fitness status score (PS score) 0;
4. Child-Pugh score A;
5. Histopathologically confirmed intrahepatic cholangiocarcinoma; consent to provide previously stored tumor tissue specimens or fresh biopsy tumor lesions;
6. unresectable ICC patients;
7. Functional indicators of vital organs meet the following requirements a Neutrophils ≥1.5*109/L; platelets≥100*109/L; hemoglobin≥9g/dl; serum albumin≥3g/dl; b Thyroid stimulating hormone (TSH) ≤ 1 times the upper limit of normal value(ULN), T3, T4 are in the normal range; c bilirubin ≤ 1.5 times ULN; Alanine aminotransferase （ALT） and Aspartate aminotransferase （AST） ≤ 1.5 times ULN; d serum creatinine ≤ 1.5 ULN, creatinine clearance rate ≥ 60ml / min;
8. The subject has at least 1 measurable liver lesion or non-liver lesion (according to RECIST 1.1);
9. Non-lactating or pregnant women, contraception during or after 3 months of treatment.

Exclusion Criteria:

1. pathological diagnosis of hepatocellular carcinoma, mixed liver cancer and other non-cholangiocarcinoma malignant tumor components;
2. patients who have received previous treatment with PD1 antibody, programmed death ligand -1 （PDL1） antibody or cytotoxic T lymphocyte-associated antigen-4 （CTLA4） antibody;
3. with other malignant tumors, except for fully treated non-melanoma skin cancer, cervical carcinoma in situ, and papillary thyroid carcinoma;
4. active tuberculosis infection. Patients with active tuberculosis infection within 1 year prior to enrollment; had a history of active tuberculosis infection more than 1 year before enrollment, did not receive formal anti-tuberculosis treatment or tuberculosis is still active;
5. Have an active, known or suspected autoimmune disease. Subjects who require only hormone replacement therapy for hypothyroidism and skin diseases that do not require systemic therapy may be enrolled;
6. previous interstitial lung disease, or (non-infectious) pneumonia and need oral or intravenous steroid therapy;
7. Long-term systemic hormones (dose equivalent to >10 mg prednisone/day) or any other form of immunosuppressive therapy are required. Subjects using inhaled or topical corticosteroids may be enrolled;
8. severe cardiopulmonary and renal dysfunction;
9. suffering from high blood pressure, and can not be well controlled by antihypertensive drugs (systolic blood pressure ≥140mmHg or diastolic blood pressure ≥90mmHg);
10. abnormal blood coagulation (PT>14s), with bleeding tendency or receiving thrombolytic or anticoagulant therapy;
11. hepatitis B virus （HBV） DNA>2000 copies/ml, hepatitis C virus （HCV） RNA>1000;
12. Significant clinically significant bleeding symptoms or a clear tendency to appear within 3 months prior to enrollment;
13. active infections requiring systemic treatment;
14. Human immunodeficiency virus (HIV) positive;
15. History of psychotropic substance abuse, alcohol abuse or drug abuse;
16. has a history of allergy to platinum;
17. Other factors that may influence the safety of the subject or the compliance of the test by the investigator. Serious illnesses (including mental illness), severe laboratory tests, or other family or social factors that require combined treatment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-05-10 (Actual); Primary Completion 2020-01-10 (Actual); Study Completion 2021-11-10 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | 12 months
  Objective response rate of advanced and unresectable intrahepatic cholangiocarcinoma in combination therapy

SECONDARY OUTCOMES:
safety: the potential side effects | 12 months
  the potential side effects
overall survival | 12 months
  From the beginning date of combined therapy to the date of death
Progression free survival | 12 months
  From the beginning date of combined therapy to the date of disease progression

CONTACTS AND LOCATIONS:
Overall Officials: Jian Zhou, MD&PhD, Principal Investigator — Fudan University
Locations (1):
- Zhongshan Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Andre T, Tournigand C, Rosmorduc O, Provent S, Maindrault-Goebel F, Avenin D, Selle F, Paye F, Hannoun L, Houry S, Gayet B, Lotz JP, de Gramont A, Louvet C; GERCOR Group. Gemcitabine combined with oxaliplatin (GEMOX) in advanced biliary tract adenocarcinoma: a GERCOR study. Ann Oncol. 2004 Sep;15(9):1339-43. doi: 10.1093/annonc/mdh351. PMID 15319238
- [Background] Kudo M, Finn RS, Qin S, Han KH, Ikeda K, Piscaglia F, Baron A, Park JW, Han G, Jassem J, Blanc JF, Vogel A, Komov D, Evans TRJ, Lopez C, Dutcus C, Guo M, Saito K, Kraljevic S, Tamai T, Ren M, Cheng AL. Lenvatinib versus sorafenib in first-line treatment of patients with unresectable hepatocellular carcinoma: a randomised phase 3 non-inferiority trial. Lancet. 2018 Mar 24;391(10126):1163-1173. doi: 10.1016/S0140-6736(18)30207-1. PMID 29433850
- [Background] El-Khoueiry AB, Sangro B, Yau T, Crocenzi TS, Kudo M, Hsu C, Kim TY, Choo SP, Trojan J, Welling TH Rd, Meyer T, Kang YK, Yeo W, Chopra A, Anderson J, Dela Cruz C, Lang L, Neely J, Tang H, Dastani HB, Melero I. Nivolumab in patients with advanced hepatocellular carcinoma (CheckMate 040): an open-label, non-comparative, phase 1/2 dose escalation and expansion trial. Lancet. 2017 Jun 24;389(10088):2492-2502. doi: 10.1016/S0140-6736(17)31046-2. Epub 2017 Apr 20. PMID 28434648
- [Derived] Shi GM, Huang XY, Wu D, Sun HC, Liang F, Ji Y, Chen Y, Yang GH, Lu JC, Meng XL, Wang XY, Sun L, Ge NL, Huang XW, Qiu SJ, Yang XR, Gao Q, He YF, Xu Y, Sun J, Ren ZG, Fan J, Zhou J. Toripalimab combined with lenvatinib and GEMOX is a promising regimen as first-line treatment for advanced intrahepatic cholangiocarcinoma: a single-center, single-arm, phase 2 study. Signal Transduct Target Ther. 2023 Mar 17;8(1):106. doi: 10.1038/s41392-023-01317-7. PMID 36928584